CLINICAL TRIAL: NCT01279395
Title: Impact of Anti-inflammatory Agents on Cholesterol Metabolism and Atherogenic Potency of Patient Plasma
Brief Title: Anti-inflammatory Agents and Cholesterol Metabolism
Status: Terminated | Type: Observational
Why Stopped: Could not recruit adequate number of subjectsa
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Allison B. Reiss, MD, Associate Professor of Medicine, Winthrop University Hospital
Other Study IDs: 151973-1
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis
Keywords: atherosclerosis; cholesterol; cyclooxygenase; gene expression; lipid metabolism
MeSH Terms: conditions — Osteoarthritis; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- naproxen: Patients age 40-70 who fulfill the American College of Rheumatology (ACR) criteria for a diagnosis of primary osteoarthritis are considered eligible. This group has been prescribed naproxen (1000 mg/day) for a minimum of two weeks.
- diclofenac: Patients age 40-70 who fulfill the ACR criteria for a diagnosis of primary osteoarthritis. The group consists of patients who have been prescribed diclofenac (150 mg/day)for a minimum of two weeks.
- celecoxib: Patients age 40-70 who fulfill the ACR criteria for a diagnosis of primary osteoarthritis are considered eligible. This group has been prescribed celecoxib (200 mg/day) for a minimum of two weeks.

SUMMARY:
We hypothesize that administration of anti-inflammatory medications such as celecoxib, naprosyn and diclofenac will cause changes in the blood plasma and white blood cells of patients such that they will be less able to efficiently process cholesterol.

DETAILED DESCRIPTION:
Drugs that inhibit cyclooxygenase (COX) are frequently administered to relieve pain and inflammation, but have been associated with cardiovascular (CV) toxicity and an elevated risk of acute myocardial infarction. We have demonstrated that drugs that inhibit the COX-2 isoform act to interfere with cellular cholesterol movement by suppressing expression of proteins that facilitate efflux of cholesterol as well as by enhancing expression of scavenger receptors that mediate cholesterol uptake. We further showed that in cultured THP-1 human macrophages, COX-2 inhibition with drugs (celecoxib, NS398) or by COX-2 RNA silencing leads to foam cell transformation, a critical component of atherogenesis. Thus, COX-2 inhibitors act in a pro-atherogenic fashion on a series of genes which we have named the "Cholesterol Metabolic Signature." Alterations in this signature may contribute to heightened risk of development of atherosclerotic CV disease associated with prolonged use of this drug class. COX enzyme activity supports cholesterol homeostasis through catalysis of prostaglandin (PG) production, and we have shown in vitro that specific subsets of these PGs (PGD2 or PGE2) are sufficient to maintain balance. The aims of this project is: In an observational study of persons with pharmacologic COX-2 selective inhibition (celecoxib) or COX-1/2 inhibition (naproxen, diclofenac), document treatment effects on the Cholesterol Metabolic Signature in isolated subject mononuclear cells and in naïve THP-1 monocytes/macrophages exposed to subject plasma. This will allow detection of variations in degree of pro-atherogenic response of the Cholesterol Metabolic Signature to COX inhibition within human patients that may be associated with a higher likelihood of developing CV sequelae. Understanding the nature of the association between COX inhibition and cholesterol metabolism, and the extent to which they may promote atherosclerotic CV disease, is of critical importance in developing analgesic and anti-inflammatory medications with a more favorable risk profile. The knowledge gained may also improve clinical decision-making by identifying subsets of patients most vulnerable to adverse CV effects of COX inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70, osteoarthritis, male or female

Exclusion Criteria:

* other known autoimmune or inflammatory rheumatic conditions, renal disease, current or recent (>1 month) corticosteroid or statin treatment, contraindications to medication (i.e. those taking oral anticoagulants, e.g. warfarin), those pregnant or trying to become pregnant or breastfeeding. Participants will not have consumed any medications containing aspirin or other NSAIDs for at least 2 weeks before the trial.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 40-70 who fulfill the ACR criteria for a diagnosis of primary osteoarthritis are considered
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-11; Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Difference in expression of the cholesterol-metabolizing enzyme cytochrome P450 cholesterol 27-hydroxylase in peripheral blood mononuclear cells (PBMC) before and after treatment with naprosyn, celecoxib or diclofenac. | 2 weeks
  PBMC are isolated directly from patient blood by Ficoll hypaque gradient centrifugation. Total RNA is obtained (TriZol) from PBMC. 27-hydroxylase message is quantitated by quantitative real-time polymerase chain reaction (QRT-PCR) using specific primers.

SECONDARY OUTCOMES:
Difference in expression of cholesterol 27-hydroxylase in naive THP-1 human macrophages incubated in plasma from patients obtained before and after treatment with naprosyn, diclofenac or celecoxib. | 2 weeks
  Comparison of abundance of the cholesterol-metabolizing enzyme cytochrome P450 cholesterol 27-hydroxylase in the THP-1 human monocyte/macrophage cell line incubated in plasma taken from the same patient before and after treatment with naprosyn, celecoxib or diclofenac. 27-hydroxylase message is quantitated by QRT-PCR and protein by immunoblot.

CONTACTS AND LOCATIONS:
Overall Officials: Allison B Reiss, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Anwar K, Voloshyna I, Littlefield MJ, Carsons SE, Wirkowski PA, Jaber NL, Sohn A, Eapen S, Reiss AB. COX-2 inhibition and inhibition of cytosolic phospholipase A2 increase CD36 expression and foam cell formation in THP-1 cells. Lipids. 2011 Feb;46(2):131-42. doi: 10.1007/s11745-010-3502-4. Epub 2010 Dec 22. PMID 21181286
- [Background] Reiss AB, Anwar F, Chan ES, Anwar K. Disruption of cholesterol efflux by coxib medications and inflammatory processes: link to increased cardiovascular risk. J Investig Med. 2009 Aug;57(6):695-702. doi: 10.2310/JIM.0b013e31819ec3c7. PMID 19289972
- [Background] Chan ES, Zhang H, Fernandez P, Edelman SD, Pillinger MH, Ragolia L, Palaia T, Carsons S, Reiss AB. Effect of cyclooxygenase inhibition on cholesterol efflux proteins and atheromatous foam cell transformation in THP-1 human macrophages: a possible mechanism for increased cardiovascular risk. Arthritis Res Ther. 2007;9(1):R4. doi: 10.1186/ar2109. PMID 17244362